CLINICAL TRIAL: NCT00927017
Title: Lakritsin Vaikutus Kaliumpitoisuuteen
Brief Title: The Effect of Liquorice on Plasma Potassium
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: When 9 subjects of targeted 12 subjects had been studied, no changes in plasma potassium were detected and it was deemed futile to continue with enrolment.
Sponsor: University of Oulu (Other)
Responsible Party: Janne Hukkanen, Oulu University Hospital, Department of Internal Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Lakritsi-2
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Glycyrrhiza glabra extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liquorice 66 g/day (Active Comparator): Liquorice given 66 grams per day for two weeks
  Interventions: Other: Liquorice 66 g/day
- Liquorice 102 g/day (Active Comparator): Liquorice given 102 grams per day for two weeks
  Interventions: Other: Liquorice 102 g/day

INTERVENTIONS:
Other: Liquorice 66 g/day — Liquorice 66 g/day for two weeks
  Other Names: Pepe Original liquorice
  Arms: Liquorice 66 g/day
Other: Liquorice 102 g/day — Liquorice 102 g/day for two weeks
  Other Names: Pepe Original liquorice
  Arms: Liquorice 102 g/day

SUMMARY:
The hypothesis is that liquorice lowers plasma potassium. This study aims to elucidate the dose-response of this effect with two doses of liquorice (66 grams or 102 grams) per day for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* age 18-40

Exclusion Criteria:

* any continuous medication
* hypertension or hypotension
* allergy to liquorice
* pregnancy or lactation
* difficult venipuncture
* drug or alcohol abuse
* participation in pharmaceutical trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in plasma potassium | 1 week, 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janne Hukkanen, MD, PhD, Principal Investigator — Oulu University Hospital, Department of Internal Medicine
Locations (1):
- Oulu University Hospital, Oulu, Finland